CLINICAL TRIAL: NCT06119802
Title: Prediction of UA/SOD Ratio as a Biomarker of Oxidative Stress in Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yinglong Hou (Other)
Responsible Party: Sponsor-Investigator, Yinglong Hou, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023(044)
Record Dates: First submitted 2023-09-06; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation; Hyperuricemia
Keywords: hyperuricemia; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Hyperuricemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atrial Fibrillation cohort: The diagnosis of AF was based on 12-lead electrocardiography (ECG) or 24-hour Holter monitoring, and classification was based on the published 2020 ESC guidelines for the diagnosis and management of AF. The exclusion criteria were as follows: (1) acute heart failure and acute myocardial infarction; (2) severe liver or kidney dysfunction (with aspartate aminotransferase or alanine aminotransferase levels three times higher than normal and estimated glomerular filtration rate <30 ml/ (min*1.73 m2)); (3) malignant tumors; and (4) missing data of laboratory indicators at baseline.
  Interventions: Diagnostic Test: atrial fibrillation
- Non-atrial Fibrillation cohort: Patients attending the Department of Cardiology to rule out atrial fibrillation.The exclusion criteria were as follows: (1) acute heart failure and acute myocardial infarction; (2) severe liver or kidney dysfunction (with aspartate aminotransferase or alanine aminotransferase levels three times higher than normal and estimated glomerular filtration rate <30 ml/ (min*1.73 m2)); (3) malignant tumors; and (4) missing data of laboratory indicators at baseline.

INTERVENTIONS:
Diagnostic Test: atrial fibrillation — ECG of atrial fibrillation last more than 30 seconds.
  Groups: Atrial Fibrillation cohort

SUMMARY:
To clarify the predictive effects of uric acid and superoxide dismutase as biomarkers of oxidative stress on atrial fibrillation, and to provide greater value for the diagnosis and prediction of atrial fibrillation. It provides a new idea for the prevention and treatment of atrial fibrillation.

DETAILED DESCRIPTION:
In recent years, a growing number of reports have shown the importance of oxidative stress in the pathophysiological mechanism of AF. During oxidative stress, there is an imbalance between the production of pro-oxidant reactive species and the antioxidant defenses of the cell, and excessive oxidation leads to oxidative damage and cell death. Redox processes can lead to atrial fibrosis and cardiac remodeling , suggesting that strategies to address myocardial oxidative stress may constitute a reasonable approach for the treatment of AF. However, few studies have reported the relationship between comprehensive oxidative stress-related biomarkers and AF. The purpose of this study was to illuminate the relationship of several blood markers of oxidative stress with AF and to provide new clues for the prevention and treatment of AF.

ELIGIBILITY:
Inclusion Criteria: This retrospective study enrolled all hospitalized patients from January 2018 to December 2020 at the Department of Cardiology in The First Affiliated Hospital of Shandong First Medical University. The diagnosis of AF was based on 12-lead electrocardiography (ECG) or 24-hour Holter monitoring, and classification was based on the published 2020 ESC guidelines for the diagnosis and management of AF.

Exclusion Criteria:

1. acute heart failure and acute myocardial infarction;
2. severe liver or kidney dysfunction (with aspartate aminotransferase or alanine aminotransferase levels three times higher than normal and estimated glomerular filtration rate <30 ml/ (min*1.73 m2));
3. malignant tumors;
4. missing data of laboratory indicators at baseline.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This retrospective study enrolled all hospitalized patients from January 2018 to December 2020 at the Department of Cardiology in The First Affiliated Hospital of Shandong First Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Uric acid/SOD ratio is associated with atrial fibrillation | 3 years
  Uric acid/SOD ratio is associated with atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Hui Tian, PhD, Study Chair — Qianfoshan Hospital
Locations (1):
- Shandong provincal Qianfoshan hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No